CLINICAL TRIAL: NCT02006420
Title: Acoustic Radiation Force Impulse/Shear Wave Velocity Imaging of the Skin in Scleroderma and Other Rheumatologic Diseases
Brief Title: Scleroderma ARFI Imaging of the Skin
Acronym: ARFI
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Dinesh Khanna, MD, MS, Principal Investigator, University of Michigan
Other Study IDs: HUM00074229
Record Dates: First submitted 2013-11-26; First posted 2013-12-10 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ARFI-SVI Ultrasound: Ultrasound imaging of forearm and thigh, lasting approximately 5-10 minutes.
  Interventions: Device: ARFI-SVI Ultrasound
- Healthy Volunteers: ARFI/SVI Ultrasound: Ultrasound imaging of forearm and thigh, lasting approximately 5-10 minutes.
  Interventions: Device: ARFI-SVI Ultrasound

INTERVENTIONS:
Device: ARFI-SVI Ultrasound — Ultrasound imaging of arm and leg lasting approximately 5-10 minutes. Participants will also undergo durometer scoring on the forearm and thigh as part of the study. This lasts approximately 5-10 minutes.

SUMMARY:
Scleroderma and other rheumatologic conditions can affect the skin. Scleroderma in particular involves skin thickening and hardening.

Currently, looking at the degree that the skin is affected by scleroderma is measured based on a combination of a physical exam and a skin biopsy.

The researchers propose to measure skin hardness using ultrasound imaging of elasticity. They will use a technique using acoustic radiation force impulse/shear wave velocity imaging , known as ARFI/SVI).

The investigators hypothesize that ARFI/SVI may be able to distinguish between normal skin and skin affected by scleroderma.. This tool may also help to quantify the amount of fibrosis in the skin.

This type of radiologic biomarker could be used to help confirm the diagnosis of scleroderma.

DETAILED DESCRIPTION:
Scleroderma as well as numerous other rheumatologic conditions can affect the skin. Scleroderma in particular causes skin thickening and hardening.

Currently, evaluation of degree to which skin is affected by scleroderma is measured by a combination of a physical exam and skin biopsy results.

The investigators propose to measure skin hardness using ultrasound elasticity imaging, in the form of acoustic radiation force impulse/shear wave velocity imaging (ARFI/SVI).

The investigators hypothesize that ARFI/SVI may be able to distinguish normal skin from skin affected by scleroderma (and other rheumatologic conditions). And, this ultrasound technique might measure the amount of fibrosis in the dermis (skin).

Such a radiologic biomarker could be used to help confirm the diagnosis of scleroderma. In addition, it may be usable for following patients over time and measuring their response to therapy and progression of disease.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Rheumatologic disease of the skin including: Limited Scleroderma, Diffuse Scleroderma, or Eosinophilic Fascitis (Schulman's Syndrome)

Exclusion Criteria:

1. None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are people aged 18 or over who are either healthy or who have scleroderma or another rheumatological condition.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Scleroderma: Scleroderma participants could have limited or diffuse scleroderma Ultrasound imaging of arm and leg lasting approximately 5-10 minutes. Participants will also undergo durometer scoring on the forearm and thigh as part of the study. This lasts approximately 5-10 minutes.
- Control: Ultrasound imaging of arm and leg lasting approximately 5-10 minutes. Participants will also undergo durometer scoring on the forearm and thigh as part of the study. This lasts approximately 5-10 minutes.
Period: Overall Study
Arm/Group | Scleroderma | Control
Started | 24 | 21
Completed | 24 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Scleroderma; Control: Ultrasound imaging of forearm and thigh, lasting approximately 5-10 minutes.
  ARFI-SVI Ultrasound: Ultrasound imaging of arm and leg lasting approximately 5-10 minutes. Participants will also undergo durometer scoring on the forearm and thigh as part of the study. This lasts approximately 5-10 minutes.
- Total: Total of all reporting groups
Arm/Group | Scleroderma | Control | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (14.6) | 47.7 (14.68) | 48.2 (14.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Skin Stiffness
Description: Skin stiffness was measured from the forearm and thigh of patients with scleroderma using ultrasound shear wave velocity imaging. Shear wave velocity is measured in meters per second (m/s).
Time Frame: Cross-sectional study, 1 visit, <1 hr
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- Scleroderma: Scleroderma participants could have limited or diffuse scleroderma. Ultrasound imaging of arm and leg lasting approximately 5-10 minutes. Participants will also undergo durometer scoring on the forearm and thigh as part of the study. This lasts approximately 5-10 minutes.
Arm/Group | Scleroderma | Control
Number analyzed (Participants) | 24 | 21
meters per second
  Forearm | 2.68 (0.82) | 2.07 (0.25)
  Thigh | 2.23 (0.48) | 2.27 (0.36)
Statistical Analysis 1: Comparison: Scleroderma vs Control; This is the p value for the mean skin thickness of the forearm; Test type: Superiority; p = 0.005, t-test, 2 sided; Unequal variance assumption
Statistical Analysis 2: Comparison: Scleroderma vs Control; This is the p value for the mean skin stiffness of the thigh; Test type: Superiority; p = 0.71, t-test, 2 sided; Unequal variance assumption

2. Secondary Outcome: Mean Skin Stiffness as Measured by Durometer Scoring
Description: Durometer scoring of skin stiffness in two groups of patients (controls and scleroderma). Durometer measurements are expressed in standardized international durometer units ranging from 0 to 100 where 100 is harder (worse outcome) The Rex Gauge model DD-3 was used. For further reference see Arthritis and Rheumatism (Arthritis Care & Research) Vol. 55. No. 4, August 15, 2006, pp. 603-609. DOI 10.1002/art.22093.
Time Frame: Cross-sectional study, 1 visit, <1 hr
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Scleroderma: Scleroderma Arm. Patients could have limited or diffuse scleroderma.Participants undergo durometer scoring on the forearm and thigh as part of the study.
- Control Arm: Healthy volunteers who do not have scleroderma.Participants undergo durometer scoring on the forearm and thigh as part of the study.
Arm/Group | Scleroderma | Control Arm
Number analyzed (Participants) | 24 | 21
units on a scale
  Forearm | 30.5 (9.4) | 19.1 (2.8)
  Thigh | 30.1 (8.5) | 19.3 (3.5)
Statistical Analysis 1: Comparison: Scleroderma; This is the p-value for the forearm; Test type: Superiority; p = 0.002, Pearson correlation
Statistical Analysis 2: Comparison: Scleroderma; This is the p-value for the thigh; Test type: Superiority; p = 0.007, Pearson correlation

3. Secondary Outcome: Linear Relationship Between Ultrasound Skin Stiffness and Durometer
Description: Pearson correlation assesses the linear relationship between Ultrasound skin stiffness measurements and Durometer scoring of skin stiffness.
  Data was combined for scleroderma and control subjects to assess the relationship and association across a broad range of skin conditions.
Time Frame: Cross-sectional study, 1 visit, <1 hr
Measure: Number; unit: Correlation coefficient
Groups:
- All Participants: Scleroderma and Healthy Volunteers
Arm/Group | All Participants
Number analyzed (Participants) | 45
Correlation coefficient
  Forearm | 0.45
  Thigh | 0.40
Statistical Analysis 1: Comparison: All Participants; This is the p value for the forearm; Test type: Superiority; p = 0.002, Pearson correlation
Statistical Analysis 2: Comparison: All Participants; This is the p value for the thigh; Test type: Superiority; p = 0.007, Pearson correlation

4. Secondary Outcome: Mean Landmark Scores
Description: Mean Landmark scores are on a scale of 0 to 3, 0 = normal and 3 =marked skin hardening.
Time Frame: Cross-sectional study, 1 visit, <1 hr
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Scleroderma | Control Arm
Number analyzed (Participants) | 24 | 21
units on a scale
  Forearm | 0.6667 [0 to 2] | 0 [0 to 0]
  Thigh | 0.58333 [0 to 2] | 0 [0 to 0]

5. Secondary Outcome: Linear Relationship Between Ultrasound Skin Stiffness and Landmark
Description: Pearson correlation assesses the linear relationship between ultrasound skin stiffness and subjective skin scoring (Landmark) of skin stiffness in all patients (controls plus scleroderma). Data was combined for scleroderma and control subjects to assess the relationship and association across a broad range of skin conditions.
Time Frame: Cross-sectional study, 1 visit, <1 hr
Measure: Number; unit: correlation coefficient
Groups:
- Stiffness vs. Landmark: Scleroderma and Healthy Volunteers
Arm/Group | Stiffness vs. Landmark
Number analyzed (Participants) | 45
correlation coefficient
  Forearm | .65
  Thigh | .55
Statistical Analysis 1: Comparison: Stiffness vs. Landmark; This is the p-value for the forearm; Test type: Superiority; p < .0001, Pearson correlation
Statistical Analysis 2: Comparison: Stiffness vs. Landmark; This is the p-value for the thigh; Test type: Superiority; p < 0.0001, Pearson correlation

6. Secondary Outcome: MRSS Scores for Scleroderma Participants.
Description: MRSS scores exist on a scale from 0 to 51 based on scores of 0 to 3 measured in 17 locations on the body, where 0 represents overall healthy skin and 51 would be the worst outcome in all 17 locations.
  MRSS measures are not taken on healthy participants.
Time Frame: Cross-sectional study, 1 visit, <1 hr
Population: Of 24 scleroderma participants, data was not available for 2.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Scleroderma Participants: Scleroderma Participants only
Arm/Group | Scleroderma Participants
Number analyzed (Participants) | 22
units on a scale | 11.27273 [2 to 29]

7. Secondary Outcome: Linear Relationship Between Ultrasound Skin Stiffness and MRSS
Description: Pearson correlation assesses the linear relationships between ultrasound skin stiffness and subjective skin scoring (MRSS) of skin stiffness. MRSS is the Modified Rodnan Score. Skin thickness is measured by clinical palpation using a 0-3 scale. 0 = normal skin; 1 = mild thickness; 2 = moderate thickness; 3 = severe thickness with inability to pinch the skin into a fold.
  Because MRSS measurements were not taken for healthy participants, no correlations are provided for them. Therefore, the correlations are based on a skin stiffness and skin scoring solely for scleroderma participants.
Time Frame: Cross-sectional study, 1 visit, <1 hr
Population: Data for 2 of 24 participants is not available.
Measure: Number; unit: correlation coefficient
Groups:
- Stiffness vs. MRSS: Scleroderma Participants only
Arm/Group | Stiffness vs. MRSS
Number analyzed (Participants) | 22
correlation coefficient
  Forearm | 0.53
  Thigh | 0.36
Statistical Analysis 1: Comparison: Stiffness vs. MRSS; This is the p-value for the forearm; Test type: Superiority; p = 0.01, Pearson correlation
Statistical Analysis 2: Comparison: Stiffness vs. MRSS; This is the p-value for the thigh; Test type: Superiority; p = 0.10, Pearson correlation

ADVERSE EVENTS:
Time Frame: single visit; less than 1 hour; no specific follow up.
Arm/Group | Scleroderma | Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes